CLINICAL TRIAL: NCT06101550
Title: A Comparative Evaluation of Partial Versus Complete Pulpotomy in Immature Young Permanent Molars Using Well-Root PT: Randomized Controlled Trial.
Brief Title: Evaluation of Partial Versus Complete Pulpotomy in Carious Immature Molars Permanent Teeth Using Bioceramic Material
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Abdel Azim, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14422023560059
Record Dates: First submitted 2023-10-18; First posted 2023-10-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Carious Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- partial pulpotomy in immature permanent teeth (Experimental): partial removal of coronal pulp tissue
  Interventions: Procedure: partial pulpotomy
- complete pulpotomy in immature permanent teeth (Active Comparator): complete removal of pulp in pulp chamber
  Interventions: Procedure: Complete pulpotomy

INTERVENTIONS:
Procedure: partial pulpotomy — Partial removal of pulp tissue in young permanent teeth
  Arms: partial pulpotomy in immature permanent teeth
Procedure: Complete pulpotomy — Complete removal of pulp tissue in young permanent teeth
  Arms: complete pulpotomy in immature permanent teeth

SUMMARY:
One of our major concerns and daily challenges is the management of carious immature permanent teeth, also known as young permanent teeth while preserving the vitality of the dental. Preserving radicular pulp tissue in these teeth allows continuing apical maturation and apical closure.

Diagnosis and treatment of carious immature permanent molars are considered a challenging aspect of daily clinical routine, where constant irritation of the pulp without treatment leads to irreversible pulpitis and necrosis, which impedes the natural root development and its complete formation ; leading at the end to a decision of extracting the tooth .Therefore; when treating immature permanent teeth, the main goal is to preserve the vitality of the pulp to guarantee natural root development.

Pulpotomy is a commonly employed treatment for this procedure involving either the removal of only the outer layer of damaged and hyperemic tissue in exposed pulps (partial pulpotomy or Cvek pulpotomy); which is a procedure staged between pulp capping and complete pulpotomy.

Complete pulpotomy is the total removal of coronal pulp tissue and the placement of a wound dressing on the canal orifice. Followed by the placement of a biocompatible material to promote healing and regeneration of the remaining vital pulp tissue.

In many studies, MTA showed high success rates in treatment of carious immature permanent molars. However, MTA is expensive and has poor handling characteristics, a long setting time and no predictable antimicrobial activity.

Recently, new bioceramics have emerged as promising materials, showing good potential for vital pulp therapy in immature permanent teeth due to their biocompatibility and favorable clinical outcomes.

Both MTA and bioceramics have almost similar compositions, but bioceramics materials contain titanium oxide and calcium phosphate, in addition to the absence of aluminum in its composition. Besides, bioceramics can release a high percentage of calcium ions early while maintaining this high percentage for 28 days, in contrast to the mineral trioxide, which showed a lower ability to release calcium ions more slowly.

Therefore, this study will be conducted to compare the effectiveness bioceramic material in partial and complete pulpotomy of immature permanent molars.

DETAILED DESCRIPTION:
comparing the effectiveness of bioceramic material in partial and complete pulpotomy in carious immature permanent molars.

ELIGIBILITY:
Inclusion Criteria:

1. Children with vital immature mandibular first permanent molars; with clinical carious exposure of the pulp and presence of bleeding upon exposure.
2. Age ranges from 6-10 years.
3. No history of spontaneous pain.
4. Absence of sinus tract, sinus swelling.
5. The posterior teeth could be restored.

Exclusion Criteria:

1-History of spontaneous pain, or pain that wakes up the child at night. 2-Teeth with closed apex. 3-Teeth with furcation, prominent radiolucency in the periapical region. 4-Teeth with excessive mobility. 5-Non-restorable molars.

-

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
post operative pain | 3 months,6 months, 1 year
  patient will be asked if there is pain or no

SECONDARY OUTCOMES:
radiographic evaluation | 3 months,6 months, 1 year
  the radiograph will be evaluated for thickening of dentine walls, root completion.